CLINICAL TRIAL: NCT05799079
Title: Phase 2 Study of Decitabine and Cedazuridine in Combination With Venetoclax for AML Relapse After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Decitabine and Cedazuridine in Combination With Venetoclax for the Treatment of Patients Who Have Relapsed Acute Myeloid Leukemia After Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to lack of accrual and loss of funding.
Sponsor: Sanjay Mohan (Other)
Collaborators: National Comprehensive Cancer Network (Network); Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sanjay Mohan, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCHEM2163
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Decitabine; cedazuridine; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Venetoclax, DEC-C) (Experimental): Patients receive venetoclax PO daily for 28 days in a 28-day cycle. Patients receive DEC-C PO daily on days 1-5 of a 28-day cycle. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.
  Interventions: Drug: Venetoclax; Drug: Decitabine; Drug: Cedazuridine; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Venetoclax — Given by mouth
Drug: Decitabine — Given by mouth
Drug: Cedazuridine — Given by mouth
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase II trial tests how well decitabine and cedazuridine (DEC-C) works in combination with venetoclax in treating acute myeloid leukemia (AML) in patients whose AML has come back after a period of improvement (relapse) after a donor stem cell transplant. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving DEC-C in combination with venetoclax may kill more cancer cells in patients with relapsed AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effect of DEC-C/venetoclax on the investigator-assessed composite complete remission (CR) rate (CR/complete remission with partial hematologic recovery [CRh]/complete remission with incomplete hematologic recovery [CRi]).

SECONDARY OBJECTIVES:

I. To assess the rate of partial response (PR) and morphologic leukemia free state (MLFS) following treatment with DEC-C/venetoclax. II. To assess the relapse free survival of patients treated with DEC-C/venetoclax.

III. To assess overall survival of patients treated with DEC-C/venetoclax. IV. To assess the safety and tolerability of DEC-C/venetoclax in the post-hematopoietic cell transplant (HCT) setting.

V. To assess the rates of measurable residual disease negativity in patients achieving a CR.

OUTLINE:

Patients receive venetoclax orally (PO) daily for 28 days in a 28-day cycle. Patients receive DEC-C PO daily on days 1-5 of a 28-day cycle. Patients undergo bone marrow biopsy and aspiration and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of signing the Informed Consent Form (ICF); must voluntarily sign an ICF and meet all study requirements
* History of morphologically confirmed AML (per World Health Organization [WHO] diagnostic criteria) with evidence of disease recurrence (>= 5% blasts consistent with prior disease) that occurs after allogeneic hematopoietic cell transplantation (HCT). Patients transplanted for another indication (e.g., myelodysplastic syndrome/chronic myelomonocytic leukemia [MDS/CMML]) who relapse with AML are eligible to enroll
* White blood cells (WBC) must be less than 25,000/ul for at least three days prior to cycle 1, day 1 (C1D1) (hydroxyurea allowed)
* A bone marrow biopsy must be performed and tissue collected for entrance to the trial
* Eastern Cooperative Oncology Group Performance Status of 0 - 2
* Alanine transaminase (ALT) serum glutamic pyruvic transaminase (SGPT) and/or aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) less than or equal to 3x upper limit of normal (ULN)
* Total bilirubin < 1.5 x ULN

  * Patients with Gilbert's syndrome (hereditary indirect hyperbilirubinemia) must have a total bilirubin of < 3 x ULN
* Calculated creatinine clearance >= 30 ml/min (per the Cockroft-Gault formula)
* Willingness to abide by all study requirements, including contraception, maintenance of a pill diary, and acceptance of recommended supportive care medications

Exclusion Criteria:

* Prior relapse or progression while receiving venetoclax or other commercially available or investigational BCL-2 inhibitor
* Anticancer therapy, including investigational agents =< 2 weeks or =< 5 half-lives of the drug, whichever is shorter, prior to C1D1. (Use of hydroxyurea is permitted)
* Inadequate recovery from toxicity attributed to prior anti-cancer therapy to =< Grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version [v]5.0), excluding alopecia or fatigue
* History of allogeneic HCT, or other cellular therapy product, within 3 months of signing consent
* Clinically active acute or chronic graft versus host disease (GVHD). Patients must be off calcineurin inhibitors for at least 4 weeks to be eligible
* Radiation therapy or major surgery within 3 weeks of signing consent
* Active, uncontrolled infection. Patients with infection under active treatment and controlled with antibiotics are eligible. Prophylaxis is acceptable
* Inability to tolerate oral medication, presence of poorly controlled gastrointestinal disease, or dysfunction that could affect study drug absorption
* Active documented central nervous system leukemia
* Concurrent treatment with a non-permitted concomitant medication
* Other malignancy IF currently being treated or likely to be treated in next 6 months except for basal or squamous cell carcinoma of the skin or cervical carcinoma in situ
* Pregnancy or breastfeeding females
* Known chronic alcohol or drug abuse
* Clinically significant cardiovascular disease with major event or cardiac intervention within the past 6 months (e.g. percutaneous intervention, coronary artery bypass graft, documented cardiac heart failure) as determined by the investigator
* Any other condition deemed by the investigator to make the patient a poor candidate for clinical trial and/or treatment with investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mohan, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: DEC-C 100mg/35mg D1-5 Venetoclax 400 mg per day (continuous)
- Dose Level -1: DEC-C 100mg/35mg D1-4 Venetoclax 400 mg per day (continuous)
- Dose Level -2: DEC-C 100mg/35mg D1-4 Venetoclax 400 mg per day (D1-21 per cycle)
- Phase 2 Expansion: Treatment dose determined from Dose De-escalation Phase
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -2 | Phase 2 Expansion
Started | 1 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated early by the funder due to slow accrual.
Arm/Group | Dose Level 1
Number analyzed (Participants) | 1
Age, Continuous [Median (Standard Deviation); unit: years] | 68 (NA) — Only 1 patient was enrolled in this cohort before the study was terminated by the funder. The standard deviation is not computable for 1 value.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved a Complete Response to Therapy
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Participants That Achieved a Partial Response to Therapy
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Rate of Morphologic Leukemia Free State (MLFS) Following Treatment With DEC-C/Venetoclax
Time Frame: Up to 24 months post-treatment.
Population: Data not collected for this outcome measure as study was terminated early.
Measure: Number; unit: participants
Arm/Group | Dose Level 1
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Relapse Free Survival
Description: Relapse free survival was estimated by the Kaplan-Meier Method
Time Frame: Up to 24 months post-treatment.
Population: Data not collected for this outcome measure as study was terminated early.
Measure: Number
Arm/Group | Dose Level 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Overall Survival
Description: Overall survival was estimated using the Kaplan-Meier method.
Time Frame: Up to 24 months post-treatment.
Population: Data not collected for this outcome measure as study was terminated early.
Measure: Number
Arm/Group | Dose Level 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Treatment-related Adverse Events
Description: List of adverse events that were attributed as related to study treatment is reported. All occurrences of a particular adverse event is reported.
Time Frame: The one patient that was enrolled on the study was on treatment for 3 months and adverse event data were followed during treatment and 35 days after completing treatment.
Measure: Number; unit: adverse events of dehydration
Arm/Group | Dose Level 1
Number analyzed (Participants) | 1
adverse events of dehydration | 5

7. Secondary Outcome: Rate of Measurable Residual Disease Negativity in Patients Achieving a CR
Time Frame: Up to 24 months post-treatment.
Population: Data not collected for this outcome measure as study was terminated early.
Measure: Number
Arm/Group | Dose Level 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The one patient that was enrolled on the study was on treatment for 3 months and adverse event data were followed during treatment and 35 days after completing treatment.
Arm/Group | Dose Level 1
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (12)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (4)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (5)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (7)
Lymphocyte count decreased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (22)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (4)
White blood cell decreased (Investigations) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT05799079/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT05799079/ICF_000.pdf